CLINICAL TRIAL: NCT06235697
Title: Androgen Suppression Combined With Elective Nodal Irradiation and Dose Escalated Prostate Treatment: A Non-Inferiority, Phase III Randomized Controlled Trial of Stereotactic Body Radiation Therapy Versus Brachytherapy Boost in Patients With Unfavourable Risk Localized Prostate Cancer
Brief Title: Androgen Suppression Combined With Nodal Irradiation and Dose Escalated Prostate Treatment
Acronym: ASCENDE-SBRT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTG-PR24; NCI-2023-09091 (Other: NCI CTRP); CCTG-PR24 (Other: NCI/CTEP)
Record Dates: First submitted 2024-01-19; First posted 2024-02-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EBRT + Brachy Boost (Active Comparator)
  Interventions: Radiation: Radiation; Drug: ADT
- SBRT (Experimental)
  Interventions: Radiation: Radiation SBRT only

INTERVENTIONS:
Radiation: Radiation — 46Gy / 23 fractions of EBRT to pelvis and prostate + LDR or HDR boost to prostate OR 25Gy / 5 fractions of EBRT to pelvis and prostate (ultrahypofractionation EBRT (SBRT)) + LDR or HDR boost to prostate.
  + Adjuvant ADT: Unfavourable Intermediate Risk: 6 months or High / Very High Risk: 24 months
  Arms: EBRT + Brachy Boost
Radiation: Radiation SBRT only — 25Gy / 5 fractions to pelvis + 40 Gy / 5 fractions to prostate (SBRT) (ultrahypofractionation EBRT (SBRT))
  Arms: SBRT
Drug: ADT — Assigned at enrollment
  Other Names: Androgen Deprivation Therapy
  Arms: EBRT + Brachy Boost

SUMMARY:
This study is being done to answer the following question: Is the strategy to give higher doses of radiotherapy treatment over a shorter period of time using special equipment and fewer treatments (also known as Stereotactic Body Radiation Therapy or SBRT) as effective as usual external radiation therapy given with a brachytherapy boost (which involves radiation sources inserted directly into the prostate)?

DETAILED DESCRIPTION:
The usual approach for patients with unfavourable prostate cancer who are not in a study is treatment with external beam radiation therapy (EBRT) to the pelvis and prostate in combination with hormone therapy (androgen deprivation therapy - ADT). To improve control of prostate cancer at risk of returning, additional treatment with a brachytherapy boost (insertion of radiation sources directly into the prostate) is recommended. For patients who get the usual approach for this cancer, about 89 out of 100 are free of cancer after 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate diagnosed within the last 9 months
* Participants with unfavourable risk prostate cancer are eligible according to the following NCCN classification guidelines (Version 4.2022 - May 10, 2022):

  • Unfavourable-intermediate risk - has one or more of the following:
* 2 or 3 Intermediate Risk Factors (IRFs): cT2b-cT2c, Gleason 7 (grade group 2 or 3), and/or PSA 10-20 ng/ml;
* Gleason 4+3 (grade group 3)
* > 50% biopsy cores positive

  • High risk - has one of the following:
* cT3a
* Gleason 8-10 (grade group 4 or 5)
* PSA > 20 ng/ml

  • Very-high risk - has at least one of the following:
* cT3b-cT4
* Primary Gleason pattern 5
* 2 or 3 high risk features: cT3a, Gleason 8-10 (grade group 4 or 5), and/or PSA > 20 ng/ml
* > 4 cores with Gleason 8-10 (grade group 4 or 5)
* ECOG performance status of 0, 1 or 2
* Participants must be ≥ 18 years of age
* Judged to be medically fit for brachytherapy
* Participant is able (i.e. sufficiently fluent) and willing to complete the quality of life and/or health utility questionnaires in either English, French or Spanish
* Participants consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each participant must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Participants must be accessible for treatment and follow-up. Investigators must assure themselves the participants enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up
* In accordance with CCTG policy, protocol treatment is to begin within 12 weeks of participant enrollment
* Participants must be willing to take precautions to prevent pregnancy while on study
* ADT (LHRH agonists, antagonists, or anti-androgens) for prostate cancer is permitted for up to 30 days before study enrollment
* 5-alpha reductase inhibitors (5-ARI) are allowed, but baseline PSA will be corrected if 5-ARI use occurs within 6 months of enrollment
* Participants may NOT have received other therapies including chemotherapy, PARPi, radioligand or other investigational drugs for prostate cancer
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Urinary function defined as International Prostate Symptom Score (IPSS) < 20. Alpha blockers are allowed to treat baseline urinary function
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial

Exclusion Criteria:

* Prior pelvic radiotherapy
* Contraindication to radical prostate radiotherapy (e.g. connective tissue disease or inflammatory bowel disease)
* Anticoagulation medication (if unsafe to discontinue for gold seed insertion or brachytherapy implant) and/or prior or current bleeding diathesis
* Prior steam vaporization (Rezum), transurethral resection of the prostate (TURP), prostatectomy (simple or radical), or any ablative therapy to the prostate (cryotherapy, HIFU, TULSA, focal laser ablation, photodynamic therapy)
* Prostate volume > 60cc before start of androgen deprivation therapy
* Anatomy that would preclude precise brachytherapy implant (such as arch interference or large median lobe)
* Evidence of castrate resistance (defined as a rising PSA > 3.0 ng/ml while testosterone is < 3.0 nmol/l)
* Hip prosthesis (unilateral hip replacement is allowed if dose constrains can be reasonably achieved.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 710 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2032-10-31 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
To compare the progression-free survival (PFS) of SBRT versus conventional EBRT plus brachytherapy boost defined as time to biochemical failure, initiation of salvage therapy, local-regional recurrence, distant progression, or death | 8.6 years

SECONDARY OUTCOMES:
Safety and tolerability assessed by CTCAE v5.0 | 8.6 years
PSA response at 4 years compared using a Cochran-Mantel-Haenszel (CMH) test | 8.6 years
Metastasis-free Survival compared using the Gray's test | 8.6 years
Cause-specific Survival compared using the Gray's test | 8.6 years
Overall Survival analysed using a Cox proportional hazards model and graphically described using the Kaplan-Meier method | 8.6 years
Participant-reported outcomes using EPIC-26 questionnaire | 8.6 years
Participant-reported tolerability using PRO-CTCAE questionnaire | 8.6 years
Economic Outcomes using EQ-5D-5L | 8.6 years
  Canadian sites only
Economic Outcomes using FACIT-COST | 8.6 years
  Canadian sites only

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, Study Chair — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, ON, Canada
Locations (53):
- United States (43):
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Memorial Hospital East, Shiloh, Illinois
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- Canada (10):
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Waterloo Regional Health Network, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Trillium Health Partners - Credit Valley Hospital, Mississauga, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data may be shared once the final analysis is complete following the Canadian Cancer Trials Group Data Sharing Policy
URL: https://www.ctg.queensu.ca/docs/public/policies/DataSharingandAccessPolicy.pdf